CLINICAL TRIAL: NCT06574789
Title: Individualised Dose Optimisation of Ganciclovir in Immunocompromised Children Trial (ID-MAGIC)
Acronym: ID-MAGIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107507
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Cytomegalovirus Viraemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: standard dosing (Active Comparator): Enrolled participant will receive standard dosing of IV Ganciclovir dependent on renal function:
  * CrCl >/= 70mL/min: 5 mg/kg IV 12 hourly
  * CrCl >/= 50-69: 2.5 mg/kg/ IV 12 hourly
  * CrCl >/= 25-49: 2.5 mg/kg IV 24 hourly
  Interventions: Drug: Standard dosing of IV ganciclovir
- Intervention: individualised dosing using a web app (Active Comparator): Enrolled participant will receive a personalised dosing of IV Ganciclovir calculated using an individualised IV ganciclovir dosing app, that considers the patient's weight, creatinine level, and at a target drug exposure (AUC24 between 40-100 mg.h/L), allowing for tailored dosing based on individual pharmacokinetic parameters.
  Interventions: Drug: Personalised dosing of IV ganciclovir

INTERVENTIONS:
Drug: Standard dosing of IV ganciclovir — IV ganciclovir at standard dosing
  Arms: Control: standard dosing
Drug: Personalised dosing of IV ganciclovir — IV ganciclovir at a personalised dosing calculated using a ganciclovir dosing web app
  Arms: Intervention: individualised dosing using a web app

SUMMARY:
This study is being conducted at seven major children's hospitals in Australia and New Zealand to test a new approach for treating a virus, called cytomegalovirus in children with weakened immune systems. The researchers want to find out if using a web app to customise the dose of a medication called ganciclovir is better at clearing the virus over a six-week period compared to the standard method of giving the medication.

DETAILED DESCRIPTION:
Immunocompromised children between 1 months to 18 years with cytomegalovirus viraemia who are admitted to one of the participating sites will be enrolled into the trial if eligible (see eligibility criteria) and randomly allocated into two groups. Children in the 'control- standard dosing group' will receive standard intravenous ganciclovir treatment for cytomegalovirus viraemia at a standard dosing of at 5mg/kg IV BD. Children in the "intervention: individualised dosing using a web app group" will receive a personalised intravenous ganciclovir dose calculated using an individualised IV ganciclovir dosing app. This approach considers the patient's weight, creatinine level, and target drug exposure, allowing for tailored dosing based on individual pharmacokinetic parameters. The virological clearance by 6 weeks of the children in each of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Immunocompromised patients including transplant recipients (haematopoietic stem cell transplant (HSCT), solid organ transplant (SOT)), those receiving chemotherapy or other immunosuppression or those with a known/suspected inborn error of immunity (determined by an immunologist); and
2. Detectable clinically significant CMV viraemia and treating clinician determines that antiviral therapy is indicated.
3. Willing to partake in the trial
4. Willing/able to attend all follow up visits and capable of completing all trial assessments.
5. Legally acceptable parent/guardian capable of providing consent on the participant's behalf.
6. Treating clinician agreeable to child being enrolled in the trial.

Exclusion Criteria:

1. Current or prior CMV infection with documented genotypic resistance to GCV (UL97 and/or UL54); or
2. Severe renal impairment (defined as estimated glomerular filtration rate (eGFR) <25mL/min); or
3. Congenital CMV infection; or
4. Life expectancy of less than 7 days as determined by the treating physician; or
5. History of allergy, or adverse reaction to GCV, aciclovir or any component of the formulation; or
6. Treating clinician determines that combination antiviral therapy is indicated for CMV infection; or
7. Has received >3 days of IV GCV or foscarnet or oral valganciclovir for the treatment of CMV infection prior to enrolment; or
8. Prior enrolment in the trial; or
9. Current recipient of another investigational product used for the treatment of CMV infection, as part of a clinical trial.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who achieve CMV virological clearance by 6 weeks | 42 days
  CMV virological clearance by 6 weeks to be compared between the two treatment groups. * Virological clearance defined as two consecutives negative CMV polymerase chain reaction results, or detectable but CMV viral load is less than the lower limit of detection. Separated by at least 72 hours by 6-weeks (42 days) after randomisation.

SECONDARY OUTCOMES:
The proportion of participants who achieve CMV virological clearance before 3-weeks | 21 days
  The proportion of children who achieve virological clearance before 3-weeks (21 days) to be compared between the two treatment arms. Virological clearance defined as two consecutives negative CMV polymerase chain reaction results, or detectable but CMV viral load is less than the lower limit of detection. Separated by at least 72 hours.
The proportion of participants who develop CMV disease by 6 weeks | 42 days
  The proportion of children who develop CMV disease by 6 weeks to be compared between the two treatment groups. CMV disease assessed by the treating clinician based on signs/symptoms of disease followed by microbiological confirmation at the 6-week assessment.
Difference between treatment groups in All-cause mortality by 6 months | 6 months
  All-cause mortality by 6 months to be compared between the two treatment groups. All-cause mortality assessed by chart ± telephone review by the research team at 6-month timepoint.
The proportion of participants who develop drug resistant CMV infection by 6 months | 6 months
  The proportion of children who develop drug resistant CMV infection by 6 months to be compared between the two treatment groups. Children with refractory or further CMV infections following resolution of the initial infection will be evaluated for CMV-resistance through gene testing (UL97 and UL54).
The proportion of participants with treatment-related adverse effects (AEs) | 42 days
  The proportion of children with any treatment-related AEs to be compared between the two treatment groups. Assessed at end of treatment or at 6 weeks (whichever is later) by the treating team.
Change in Quality of Life measured over 6 months using the EQ-5D-Y Questionnaire. | 7 days, 42 days, 180 days
  Quality of Life (QoL) over the 6-month period following randomisation to be compared between the two treatment groups using the QoL EQ-5D-Y questionnaire, assessed at 7 days, 42 days and 180 days.
  The EQ-5D-Y descriptive system comprises the following five dimensions: mobility, looking after oneself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems.
  The final question measures how good or bad the participants' health is that day on a scale from 0 to 100. 100 means the best health they can imagine and 0 means the worst health they can imagine.
Difference between treatment groups in cost-effectiveness over the 6-month period following randomisation | 6 months
  The total sum of all hospital and patient/family resources required per patient over the 6-month period to be compared between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gwee, Principal Investigator — Murdoch Childrens Research Institute
Locations (7):
- Australia (6):
  - Sydney Children's Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - The Royal Children's Hospital, Melbourne, Victoria
  - Monash Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Starship Children's Hospital, Auckland, North Island, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Beginning 12 months following analysis and article publication, upon approval of the request, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access:
  * Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, and appendices)
  * Trial protocol, Statistical Analysis Plan, PICF
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months following analysis and article publication, upon approval of the request
Access Criteria: Researchers must be from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Background] Heston SM, Young RR, Tanaka JS, Jenkins K, Vinesett R, Saccoccio FM, Martin PL, Chao NJ, Kelly MS. Risk Factors for CMV Viremia and Treatment-Associated Adverse Events Among Pediatric Hematopoietic Stem Cell Transplant Recipients. Open Forum Infect Dis. 2021 Dec 16;9(2):ofab639. doi: 10.1093/ofid/ofab639. eCollection 2022 Feb. PMID 35111869
- [Background] Chan S, Godsell J, Horton M, Farchione A, Howson LJ, Margetts M, Jin C, Chatelier J, Yong M, Sasadeusz J, Douglass JA, Slade CA, Bryant VL. Case Report: Cytomegalovirus Disease Is an Under-Recognized Contributor to Morbidity and Mortality in Common Variable Immunodeficiency. Front Immunol. 2022 Feb 15;13:815193. doi: 10.3389/fimmu.2022.815193. eCollection 2022. PMID 35242131
- [Background] El Haddad L, Ghantoji SS, Park AK, Batista MV, Schelfhout J, Hachem J, Lobo Y, Jiang Y, Rondon G, Champlin R, Chemaly RF. Clinical and economic burden of pre-emptive therapy of cytomegalovirus infection in hospitalized allogeneic hematopoietic cell transplant recipients. J Med Virol. 2020 Jan;92(1):86-95. doi: 10.1002/jmv.25574. Epub 2019 Sep 3. PMID 31448830
- [Background] Singh N, Winston DJ, Razonable RR, Lyon GM, Silveira FP, Wagener MM, Limaye AP. Cost-effectiveness of Preemptive Therapy Versus Prophylaxis in a Randomized Clinical Trial for the Prevention of Cytomegalovirus Disease in Seronegative Liver Transplant Recipients With Seropositive Donors. Clin Infect Dis. 2021 Nov 2;73(9):e2739-e2745. doi: 10.1093/cid/ciaa1051. PMID 32712663
- [Background] Tan SK, Waggoner JJ, Pinsky BA. Cytomegalovirus load at treatment initiation is predictive of time to resolution of viremia and duration of therapy in hematopoietic cell transplant recipients. J Clin Virol. 2015 Aug;69:179-83. doi: 10.1016/j.jcv.2015.06.006. Epub 2015 Jun 10. PMID 26209403
- [Background] Rastogi S, Ricci A, Jin Z, Bhatia M, George D, Garvin JH, Hall M, Satwani P. Clinical and Economic Impact of Cytomegalovirus Infection among Children Undergoing Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2019 Jun;25(6):1253-1259. doi: 10.1016/j.bbmt.2018.11.028. Epub 2018 Nov 29. PMID 30502538
- [Background] Camargo JF, Kimble E, Rosa R, Shimose LA, Bueno MX, Jeyakumar N, Morris MI, Abbo LM, Simkins J, Alencar MC, Benjamin C, Wieder E, Jimenez A, Beitinjaneh A, Goodman M, Byrnes JJ, Lekakis LJ, Pereira D, Komanduri KV. Impact of Cytomegalovirus Viral Load on Probability of Spontaneous Clearance and Response to Preemptive Therapy in Allogeneic Stem Cell Transplantation Recipients. Biol Blood Marrow Transplant. 2018 Apr;24(4):806-814. doi: 10.1016/j.bbmt.2017.11.038. Epub 2017 Dec 5. PMID 29217388
- [Background] Acquier M, Taton B, Alain S, Garrigue I, Mary J, Pfirmann P, Visentin J, Hantz S, Merville P, Kaminski H, Couzi L. Cytomegalovirus DNAemia Requiring (Val)Ganciclovir Treatment for More Than 8 Weeks Is a Key Factor in the Development of Antiviral Drug Resistance. Open Forum Infect Dis. 2023 Jan 23;10(2):ofad018. doi: 10.1093/ofid/ofad018. eCollection 2023 Feb. PMID 36817745
- [Background] Jang JE, Hyun SY, Kim YD, Yoon SH, Hwang DY, Kim SJ, Kim Y, Kim JS, Cheong JW, Min YH. Risk factors for progression from cytomegalovirus viremia to cytomegalovirus disease after allogeneic hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2012 Jun;18(6):881-6. doi: 10.1016/j.bbmt.2011.10.037. Epub 2011 Nov 4. PMID 22062802
- [Background] Launay E, Theoret Y, Litalien C, Duval M, Alvarez F, Lapeyraque AL, Phan V, Larocque D, Poirier N, Lamarre V, Ovetchkine P. Pharmacokinetic profile of valganciclovir in pediatric transplant recipients. Pediatr Infect Dis J. 2012 Apr;31(4):405-7. doi: 10.1097/INF.0b013e3182463a19. PMID 22198827
- [Background] Martson AG, Edwina AE, Kim HY, Knoester M, Touw DJ, Sturkenboom MGG, Alffenaar JC. Therapeutic Drug Monitoring of Ganciclovir: Where Are We? Ther Drug Monit. 2022 Feb 1;44(1):138-147. doi: 10.1097/FTD.0000000000000925. PMID 34610621
- [Background] Franck B, Woillard JB, Theoret Y, Bittencourt H, Demers E, Briand A, Marquet P, Lapeyraque AL, Ovetchkine P, Autmizguine J. Population pharmacokinetics of ganciclovir and valganciclovir in paediatric solid organ and stem cell transplant recipients. Br J Clin Pharmacol. 2021 Aug;87(8):3105-3114. doi: 10.1111/bcp.14719. Epub 2021 Jan 19. PMID 33373493
- [Background] Moretti S, Zikos P, Van Lint MT, Tedone E, Occhini D, Gualandi F, Lamparelli T, Mordini N, Berisso G, Bregante S, Bruno B, Bacigalupo A. Forscarnet vs ganciclovir for cytomegalovirus (CMV) antigenemia after allogeneic hemopoietic stem cell transplantation (HSCT): a randomised study. Bone Marrow Transplant. 1998 Jul;22(2):175-80. doi: 10.1038/sj.bmt.1701302. PMID 9707026
- [Background] Al Yazidi LS, Mitchell R, Palasanthiran P, O'Brien TA, McMullan B. Management and prevention of cytomegalovirus infection in paediatric hematopoietic stem cell transplant (HSCT) recipients: A binational survey. Pediatr Transplant. 2019 Aug;23(5):e13458. doi: 10.1111/petr.13458. Epub 2019 May 12. PMID 31081265
- [Background] Jorga K, Reigner B, Chavanne C, Alvaro G, Frey N. Pediatric Dosing of Ganciclovir and Valganciclovir: How Model-Based Simulations Can Prevent Underexposure and Potential Treatment Failure. CPT Pharmacometrics Syst Pharmacol. 2019 Mar;8(3):167-176. doi: 10.1002/psp4.12363. Epub 2018 Dec 18. PMID 30354026
- [Background] Yong MK, Shigle TL, Kim YJ, Carpenter PA, Chemaly RF, Papanicolaou GA. American Society for Transplantation and Cellular Therapy Series: #4 - Cytomegalovirus treatment and management of resistant or refractory infections after hematopoietic cell transplantation. Transplant Cell Ther. 2021 Dec;27(12):957-967. doi: 10.1016/j.jtct.2021.09.010. Epub 2021 Sep 21. PMID 34560310
- [Background] Xia W, Li HCW, Lam KWK, Chung OKJ, Song P, Chiu SY, Chan CG, Ho KY. The Impact of Hematologic Cancer and Its Treatment on Physical Activity Level and Quality of Life Among Children in Mainland China: A Descriptive Study. Cancer Nurs. 2019 Nov/Dec;42(6):492-500. doi: 10.1097/NCC.0000000000000661. PMID 30433896
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- See also: National Ethics Advisory Committee. 2019. National Ethical Standards for Health and Disability Research and Quality Improvement. Wellington: Ministry of Health — http://neac.health.govt.nz/assets/Uploads/NEAC/publications/national-ethical-standards-health-disability-research-quality-improvement-2019.pdf